CLINICAL TRIAL: NCT04755647
Title: Safety & Efficacy of Topical Nitric Oxide Releasing Solution (NORS) Delivered as an Adjunctive Footbath Treatment as Compared to Placebo in the Management of Diabetic Foot Ulcers
Brief Title: Nitric Oxide Footbath for Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanotize Research and Development corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFU-CTP-01
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: nitric oxide; diabetic wounds; diabetic foot ulcer; drug resistent wound
MeSH Terms: conditions — Diabetic Foot | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, placebo controlled parallel group,clinical safety study comparing an investigational drug add-on to a placebo control. Up to 40 participants with mildly infected neuropathic or non-neuropathic or neuro-ischemic diabetic foot ulcers will be enrolled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Packaging will be generic, coded and indistinguishable from placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide-Releasing Solution (NORS) (Experimental): Five litre foot bath delivery NORS
  Interventions: Drug: Nitric Oxide-Releasing Solution
- Saline (Placebo Comparator): Five litre foot bath delivery NORS
  Interventions: Drug: Saline solution, hypotonic

INTERVENTIONS:
Drug: Nitric Oxide-Releasing Solution — Active antimicrobial
  Arms: Nitric Oxide-Releasing Solution (NORS)
Drug: Saline solution, hypotonic — Placebo
  Arms: Saline

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of a nitric oxide releasing solution, delivered as a footbath, to act as an antimicrobial treatment for participants presenting with a diabetic foot ulcer.

DETAILED DESCRIPTION:
It is hypothesized that a single, relatively short exposure (three times a week for a half hour) of a nitric oxide releasing solution (NORS) for four (4) week period will be well tolerated and may have other beneficial secondary outcomes for individuals presenting with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Non-hospitalized, ambulatory patients with controlled diabetes mellitus as determined by physician diagnosis recorded in the medical record. Diabetes may be treated with insulin, oral hypoglycemic agents or diet alone. Patient glycaemic control (HbA1c) should be less than or equal to 12 % within 2 weeks of enrollment;
2. Must be ≥ 19 years of age unless local laws dictate otherwise;
3. Participants must be considered reliable, willing and able to give signed informed consent, and sign the informed consent form.
4. Participant is willing to be randomized and able to comply with the protocol
5. Participants must have either:

   i) 1 or more full thickness ulcers on the foot below the malleoli with a surface area exceeding 0.5 cm2 (50 mm2) after debridement (full thickness means extending through the epidermis and dermis but not involving tendon, bone, or joint capsule); or ii) 1 or more partial thickness ulcers (i.e., do not completely penetrate the dermis) of forefoot or digits; or iii) 1 or more ulcers of the forefoot or digits have granulation tissue at their base.
6. Participants must have localized mild infection of at least 1 ulcer that would ordinarily be treated on an outpatient basis. Mild infection of an ulcer is defined by the presence of at least 2 manifestations of inflammation (purulence, erythema, pain, tenderness, warmth, or induration) which is limited to the skin or superficial subcutaneous tissues. If there is more than one ulcer meeting eligibility, the Investigator will determine which ulcer will be followed for the course of the study.
7. Mild infection defined by IDSA criteria34:

   i) "Local infection involving only the skin and the subcutaneous tissue (without involvement of deeper tissues and without systemic signs as described below).

   ii) If erythema, must be >0.5 cm to ≤2 cm around the ulcer. Exclude other causes of an inflammatory response of the skin (e.g., trauma, gout, acute Charcot neuro-osteoarthropathy, fracture, thrombosis, venous stasis)."
8. Participants who have been previously treated or are currently under treatment for a localized infection of an ulcer may be enrolled if there has been an inadequate response to treatment and the ulcer is still infected as described above.
9. Participants must have a radiograph (appropriate views as determined by the investigator) within the 2 weeks prior to entry showing no evidence of cortical destruction consistent with osteomyelitis in the affected foot.
10. Participants must have either:

    i) A palpable dorsalis pedis or posterior tibial pulse in the affected foot; or ii) If the pulse is congenitally absent or not palpable due to edema, a Dopplerable dorsalis pedis or posterior tibial pulse measured at ≥ 30 mm Hg; or iii) If there are no palpable pulses, non Dopplerable pulses, rest pain, or claudication on walking less than one block are present, the patient may be enrolled only if a vascular surgeon has determined that vascular surgery, angioplasty or amputation is not warranted.
11. Participants must have no more than a reduced wound area of ≤30% documented by the PI, during the 2 weeks of screening, in which patients received institutional standard of care (SOC)
12. Participants may not be taking or have received any other investigational therapy or approved therapy (i.e., drug or device) for investigational use within the 30 days prior to entry.
13. Female Participants must be postmenopausal for at least 6 months; surgically sterilized (hysterectomy or tubal ligation); or, if of child-bearing potential, must have a negative pregnancy test prior to entry and must be willing to use one highly effective birth control method which include: hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy and tubal ligation or to use two forms of effective birth control methods which include: barrier methods of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge). The Participants must have used the birth control method for at least 2 complete menstrual cycles prior to study entry.

Exclusion Criteria

1. Participants with limb threatening infection, extensive cellulitis (≥2 cm beyond the ulcer), lymphangitis, fasciitis, deep tissue infection, an abscess, or other evidence of local complications of infection.
2. Participants with symptoms of systemic infection (e.g., severe hyperglycemia, ketoacidosis, azotemia).
3. Participants requiring concurrent local or systemic antimicrobials during the study period for any infection, including diabetic foot ulcer.
4. Participants who are currently treated by dialysis, awaiting dialysis or who have an estimated glomerular filtration rate of ≤20 mL/min/173 m2.
5. Participants who are expected to be unable to care for their ulcer because of hospitalization, vacation, disability, etc. during the study period.
6. Participants with known active alcohol or substance abuse within the 6 months preceding study entry.
7. Participants who are receiving systemic corticosteroids (in a dose equivalent to ≥ 20 mg of prednisone per day) immunosuppressive radiation therapy, or cytotoxic agents
8. Participants who require treatment for a primary or metastatic malignancy (other than squamous or basal cell carcinoma of the skin).
9. Participants with a systemically immunocompromising disease, such as acquired immune deficiency syndrome or known human immunodeficiency virus (HIV) positivity.
10. Participants who have an unexplained fever or chills during the week prior to enrollment.
11. Participants with other conditions considered by the investigator to be reasons for disqualification that may jeopardize patient safety or interfere with the objectives of the trial (e.g., acute illness or exacerbation of chronic illness, lack of motivation, history of poor compliance).
12. Women who are breast feeding, pregnant or attempting to become pregnant.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
To measure the number of participants discontinued or lost to follow-up in the NORS compared to hypotonic saline in participants with diabetic foot ulcers (DFU) | 28 days
  Proportion of participants lost-to-follow-up, discontinuing study treatment due to intolerance or adverse events, or initiating new medications or treatments, or leaving/discontinuing the study for any other reason
To measure the severity of adverse events of NORS compared to hypotonic saline in participants with DFU | 29 days
  Severity as measured by adverse event scale (1-5) and frequency of adverse events that results in discontinuation of the investigative treatment.
To measure the negative changes in laboratory values of NORS compared to hypotonic saline with DFU | 29 days
  Proportion of negative laboratory changes resulting in discontinuation of investigative treatments.
To measure the negative changes in vital sign during NORS compared to hypotonic saline administration in participants with DFU | 29 days
  Proportion of subjects with deterioration in vital signs resulting in discontinuation of investigative treatment.
To measure worsening of wound infection during NORS compared to hypotonic saline administration in participants with DFU | 29 days
  Proportion of subjects with incidence of infection resulting in discontinuation of the investigative treatment.
To measure worsening of wound area during NORS compared to hypotonic saline administration in participants with DFU | 29 days
  Proportion of subjects with increased wound area resulting in discontinuation of the investigative treatment.
To measure the methemoglobin percent level during NORS compared to hypotonic saline administration in participants withe DFU | 29 days
  Proportion of subjects with an increase in methemoglobin percent level resulting in discontinuation of the investigative treatment.

SECONDARY OUTCOMES:
To measure the efficacy of NORS compared to placebo on the change in pathogen load in participants with DFU | 29 days
  Mean change in pathogen density as measured by colony forming units per milliliter (cfu/mL) compared to control
To measure the efficacy of NORS compared to placebo on the change in bacterial load (CFU/mL) in participants with DFU | 29 days
  Proportion of participants with a reduction in bacterial load as compared to control
To measure the efficacy of NORS compared to placebo on the reduction of the number of clinical signs of infection in participants with diabetic foot ulcers (DFU) | 29 days
  Proportion of participants with Clinical Response defined as resolution of one or more clinical signs of infection reported compared to control
To measure the efficacy of NORS compared to placebo on the change in wound bacterial microbiota (species) in participants with DFU | 29 days
  Mean changes in percentage of bacterial microbiota (species) will be determined by comparing to control
To measure the efficacy of NORS compared to placebo on the change in wound area in participants with DFU | 29 days
  Mean % change in wound area calculated for DFU compared to control

CONTACTS AND LOCATIONS:
Overall Officials: Scott Schumacher, MD, Principal Investigator — Achilles Foot Health Centre
Locations (1):
- Achilles Foot Health Centre, Vancouver, British Columbia, Canada